CLINICAL TRIAL: NCT02575053
Title: Switching to Powder Free Latex Gloves in the Entire OR as Part of a New ' Latex Safe' Protocol: a Safe Alternative? A Prospective, Observational Cohort Study
Brief Title: Safety of a Powder-free Latex Allergy Protocol in the Operating Theatre: A Prospective, Observational Cohort Study
Status: Completed | Type: Observational
Sponsor: Jessa Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 15.107/anesth15.02
Record Dates: First submitted 2015-10-06; First posted 2015-10-14 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-11

CONDITIONS: Latex Hypersensitivity; Latex Allergy
Keywords: latex allergy; latex hypersensitivity; powder free latex surgical gloves; latex safe protocol
MeSH Terms: conditions — Latex Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Latex group: patients who report ( a high risk for) latex allergy and will be operated on
  Interventions: Procedure: assessment of a new latex protocol

INTERVENTIONS:
Procedure: assessment of a new latex protocol — 1. All powdered latex surgical gloves are removed from the operating theatres, recovery room and surroundings starting from 01-07-2015 in order to create a latex safe environment.
     Steps 2 and 3 remain unchanged in respect to ASA( American Society of Anesthesiologists) protocol.
  2. Removal of all materials containing latex from the resuscitation carts.
  3. Further requirements in case of latex allergic patients:
     * Identification of patients with (suspected) latex allergy.
     * All materials used during the procedure (catheters, drains, monitoring equipment,…) should be checked for latex.
  All latex containing materials should be removed from the room and latex free alternatives should be available.
  * All staff present in the room should use latex free synthetic gloves.
  * Operating tables and supports should be made of latex free material or should be covered with blankets.
  * The entire OR staff is thoroughly educated concerning the latex safe protocol.

SUMMARY:
Study objectives

Primary objective:

This study wants to evaluate the safety of a latex safe protocol as proposed by the Australasian Society of Clinical Immunology and Allergy. In other words,the investigators hope to demonstrate that patients with known latex allergy or latex sensitisation can be treated safely in operating theatres without special requirements towards scheduling provided that all powdered latex gloves are removed from the OR environment( preparation rooms, theatres, recovery room and surroundings). In contrast, earlier guidelines require the theatre to be left unused during at least 3 hours before a patient with suspected latex allergy can be operated on in this theatre.

Secondary objectives:

* The investigators want to evaluate to what extend patients who report a latex allergy show risk factors of latex allergy.
* To investigate to what extend latex allergy was proven by laboratory testing or skin testing in patients who report a latex allergy.
* Type of latex allergic reaction when patients report a latex allergy.
* The level of satisfaction of surgeons and OR scheduling staff with the new latex safe protocol and with the switching to powder free latex gloves.

DETAILED DESCRIPTION:
Introduction

Allergic reactions to natural rubber latex( NRL, or Latex) are an important issue in daily anesthesia practice. Latex allergy may result in lesions consistent with irritation dermatitis and type 4 allergic contact dermatitis. But it may also result in type 1 allergic reactions which are potentially lethal.(1) The prevalence of latex allergy in a general population is estimated less than 1%, but sensitization can rise up to 5.4-7.6%.(3,4) In certain populations at risk, the prevalence of latex allergy and sensitization rises up to 17% in health care workers an even 73% in patients who were exposed to latex on a regular basis( eg. Patients with spina bifida).

These patients require special logistic and organizational requirements during their stay in the operating room. Nowadays, both guidelines from the Belgian Society of Anesthesiology and Resuscitation(BVAR-SARB) as the American Association of Anesthesiologists recommend these patients to be scheduled as the first case of the day.(1,3) In this way, these patients are treated in an environment with a minimal amount of airborne latex particles. After all, studies have proven that using powdered latex gloves causes a substantial contamination of the operating room. Latex particles can even remain airborne up to 5 hours afterwards.(1,3,5).

In consequence, the guidelines mentioned earlier dictate patients with a (high risk for) latex allergy to be treated in an operating theatre left unused during at least 3 to 6 hours.(1,2,6) Of course, such requirements can result in organizational problems potentially resulting in delaying procedures, financial losses, patient discomfort and dissatisfaction with both patients as well as hospital staff.

The last years, some professionals have suggested the idea that planning these patients as first case of the day is no longer necessary because of certain technical evolutions in current operating room practice.(7) In a guideline published by the Australasian Society of Clinical Immunology and Allergy (last updated March 2010), patients at risk or with known latex allergy are no longer scheduled as first case of the day. However, this requires the removal of all powdered latex gloves from the OR (including pre-anesthesia unit, operating theatres, post anesthesia care unit and surroundings).(8) The requirement for a completely latex free environment en materials when operating on a actual patient with (suspected) latex allergy remains unchanged.

Although several studies have shown the importance of powdered gloves in the spread of airborne latex particles and the basis for this protocol seams acceptable and logical, there is currently no literature confirming the safety of this practice in a clinical setting.

Study objective

Primary objective:

This study wants to evaluate the safety of a latex safe protocol as proposed by the Australasian Society of Clinical Immunology and Allergy. In other words,the investigators hope to demonstrate that patients with known latex allergy or latex sensitisation can be treated safely in operating theatres without special requirements towards scheduling provided that all powdered latex gloves are removed from the OR environment (preparation rooms, theatres, recovery room and surroundings). In contrast, earlier guidelines require the theatre to be left unused during at least 3 hours before a patient with suspected latex allergy can be operated on in this theatre.

Secondary objectives:

* The investigators want to evaluate to what extend patients who report a latex allergy show risk factors of latex allergy.
* To investigate to what extend latex allergy was proven by laboratory testing or skin testing in patients who report a latex allergy.
* Type of latex allergic reaction when patients report a latex allergy.
* The level of satisfaction of surgeons and OR scheduling staff with the new latex safe protocol and with the switching to powder free latex gloves.

Study procedure

Pre-operative setting:

Medical history, including allergies of every patient will be assessed . Every patient with (suspected) latex allergy who will undergo surgery will be approached to participate in this study. There are no restrictions regarding type of surgery.

The research team will ask all eligible patients to sign an informed consent. The researchers will ask all patients who are willing to participate to complete a short questionnaire.

Patients refusing to participate will be treated by the same protocol. However, they will not be contacted in order to provide further medical data in relation to this study.

During the stay in the OR:

Nursing staff and the anesthesiologist perform a time-out procedure prior to surgery. A (suspected) latex allergy is marked in the electronic case file. The software registers this cases and sends a confirmation to the research team.

At the end of the procedure, the anesthesiologist marks if a latex allergic reaction has occurred through a pop -up in the electronic case file.

Post-operative setting:

• Recovery room: Continuation of the latex safe protocol. When the patient is discharged to the ward, a pop-up in the electronic case file asks if any type of latex allergic reaction has occurred.

The patient receives a short note, explaining that the research team will contact him/her after 72 hours.

• Wards/ discharge from hospital: The research team will contact every patient who was marked latex allergic 72 hours after their surgery to answer the questionnaire about any allergic reaction to latex( by phone or in person).

Types of latex reactions:

1. Irritation dermatitis: a non-allergic reaction of the skin to an irritans. Lesions are limited to the area of contact and may occur minutes to hours after exposure. Symptoms include itching, erythema, a burning sensation, blistering, flakiness and fissuring of the skin. This type of reaction is never life-threatening.(1,3,6)
2. Allergic contact dermatitis or delayed cell- mediated hypersensitivity reaction or type 4 reaction: T- cell mediated sensitivity for chemical additives absorbed by the skin. Lesions occur after 6 to 48 hours following exposure and peak after 48 to 72 hours. The lesions may exceed the contact area and consist of itching, erythema, blistering or flakiness.( Symptoms often resemble those of irritation dermatitis.)(1,3,6)
3. IgE mediated immediate hypersensitivity( type 1 reaction:

Based on B-cell mediated production of IgE (immunoglobulin E) antibodies towards Hev b latex proteins after a first exposure. Symptoms already occur after a few minutes up to 1 hour, depending of the route of exposure (inhalation, parenteral or mucous membrane exposure). The severity of the reaction also varies in relation to the route of exposure. Type 1 allergic reactions in response to latex exposure may be lethal.(1,2,3)

Note:

• If the research team( or in daily practice: the attending physician) suspects a latex allergic reaction during the study period , they will determine RIA(radioimmunoassay) - tryptase in case of an anaphylactic reaction. Furthermore, the patient will be referred to an allergy consultant for skin prick test in order to confirm a possible latex allergy.

Satisfaction about the newly implemented protocol:

Starting from 01-02-2016, the research team will investigate the level of satisfaction about the newly implemented protocol by means of a short questionnaire( written or E-mail) sent to all involved surgeons and OR scheduling staff.

With this questionnaire, the investigators want to evaluate

* general satisfaction regarding the new protocol by means of a numeric rating scale ranging from 0 (very unsatisfied) up to 10 (very satisfied).
* whether this new protocol has simplified the OR schedule. The investigators will do so by means of a numeric rating scale ranging from 0 (not true at all) up to 10(absolutely true).
* the level of satisfaction regarding the new type of surgical gloves in case the surgeon had to switch.The investigators will do so by means of a numeric rating scale ranging from 0 (very unsatisfied) up to 10 (very satisfied).

ELIGIBILITY:
Inclusion Criteria:

1. All patients who report prior latex allergic reactions
2. High risk patients:

   * Frequent blather catheterization: meningomyelocoele, spina bifida, congenital defects of the uro-genital tract.
   * A medical history of multiple surgical procedures
   * Atopic constitution( asthma/hay fever/ eczema) and/ or a specific food allergy,eczema) and/ or a specific food allergy( avocado, kiwi, banana, hazelnut, stone fruit, chest nut and to a lesser extent grapes, mango, melon, pineapple, figs, cherry, passion fruit, walnut)(9)
3. professional exposure: health care workers, hairdressers, chemical industries

Exclusion Criteria:

* The patient refuses to cooperate. These patients will be treated in the same way, although we will not collect any data.
* The patient patient is unable to cooperate as a result of circumstances that may interfere with collecting the data or make them unreliable. Eg. Language barriers.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Every patient with (suspected) latex allergy who will undergo surgery will be approached to participate in this study. There are no restrictions regarding type of surgery (both inpatient and outpatient surgery)
Sampling Method: Non-Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
The number and type of latex allergic reactions occuring in our included patients up to 72 hours post-operatively. | 72 hours after surgery
  The research team wants to investigate how many latex allergic reactions occur. types:
  1. Irritation dermatitis: non-allergic reaction to an irritans,minutes to hours after exposure. Symptoms:
     itching, erythema, a burning sensation, blistering, flakiness and fissuring of the skin. Never life-threatening.
  2. Allergic contact dermatitis( type 4 reaction): T- cell mediated sensitivity for chemical additives absorbed by the skin. Occurs 6 to 48 hours following exposure and peaks after 48 to 72 hours. Lesions may exceed the contact area and consist of itching, erythema, blistering or flakiness.( cf irritation dermatitis.)
  3. IgE mediated immediate hypersensitivity( type 1 reaction):
  B-cell mediated production of IgE antibodies towards Hev b latex proteins. Symptoms: after a few minutes up to 1 hour, depending of the route of exposure( inhalation, parenteral,mucous membrane exposure). Severity also varies in relation to the route of exposure. Potentially lethal anaphylaxis.

SECONDARY OUTCOMES:
How many patients (percentage of patients) who report a latex allergy have confirmed this diagnosis by laboratory testing or skin prick tests? Assessment by questionnaire | baseline
Prevalence of risk factors of latex allergy in the study population. assessment by questionnaire | baseline
  To what extend do patients who report a latex allergy show risk factors such as:
  Congenital defects of the genito-urinary tract
  Spina bifida
  Meningomyelocoele
  a medical history consisting of multiple surgical procedures
  Food allergies (tropical fruit, nuts, stone fruit, avocado, others)
  Atopic constitution( asthma, eczema, rhinitis, hay fever)
  Professional exposure( hairdressers, health care workers, latex exposure in latex industries or chemical related jobs)
  (anaphylaxis of unknown origin during previous hospital stays or procedures)
General satisfaction. Assessment by questionnaire | Assessment 8 months after introduction of the protocol
  This study wants to evaluate the level of satisfaction with surgeons and OR scheduling staff regarding the newly implemented protocol.The investigators will do so by scoring satisfaction on numeric rating scales(NRS).The research team will evaluate:
  General satisfaction by means of a numeric rating scale ranging from 0(very dissatisfied) to 10 ( very satisfied).
  The new protocol was implemented starting from 01-07-2015. The investigators will evaluate general satisfaction 8 months after implementation( period of 01-02-2016 till 01-03-2016).
simplifacation of the OR schedule. Assesment by questionnaire | assessment up to 8 months after introduction of the protocol
  The research team will evaluate whether this new protocol has simplified the OR schedule. The investigators will do so by means of a numeric rating scale ranging from 0(not true at all) up to 10(absolutely true) which has to be answered by surgeons and OR scheduling staff.
  The investigators will evaluate this up to 8 months after introduction of the new protocol(period of 01-02-2016 till 01-03-2016).The new protocol was implemented starting from 01-07-2015.
Satisfaction regarding a new type of surgical gloves | assessment up to 8 months after introduction of the protocol
  The investigators will evaluate the level of satisfaction regarding the new type of surgical gloves in case the surgeon had to switch. We will do so by means of a numeric rating scale ranging from 0 (very unsatisfied) up to 10 (very satisfied). The investigators will evaluate this up to 8 months after introduction of the new protocol( period of 01-02-2016 till 01-03-2016).The new protocol was implemented starting from 01-07-2015.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Ory, MD, Principal Investigator — Attending, department of anesthesiology; Björn Stessel, MD, Principal Investigator — Attending, department of anesthesiology
Locations (1):
- Jessaziekenhuis Hasselt, Hasselt, Limburg, Belgium

REFERENCES:
- [Background] 1. American Society of Anesthesiologists Committee on Occupational Health of Operating Room Personnel. Natural Ruber Latex Allergy: Considerations for anesthesiologists. American Society of Anesthesiologists.[brochure] 2005: 1-30.
- [Background] 2. Association of Surgical Technologists. Guideline statements for the N atural Rubber Latex Protein allergic patient in the operating room environment(adopted BOD October 2005, updated BOD January 2014). [available from: www.ast.org] accessed 19/08/2015.
- [Background] Demaegd J, Soetens F, Herregods L. Latex allergy: a challenge for anaesthetists. Acta Anaesthesiol Belg. 2006;57(2):127-35. PMID 16916182
- [Background] Reines HD, Seifert PC. Patient safety: latex allergy. Surg Clin North Am. 2005 Dec;85(6):1329-40, xiv. doi: 10.1016/j.suc.2005.09.014. PMID 16326213
- [Background] Becker HS. An analysis of the epidemiology of latex allergy: implications for primary prevention. Medsurg Nurs. 2000 Jun;9(3):135-43. PMID 11033703
- [Background] 6. American Association of Nurse Anesthetists. Latex allergy management( Guidelines). [available from: www.aana.org] accessed 15/08/2015.
- [Background] Sleth JC. [Starting the day with latex-sensitised patients: still up to date?]. Ann Fr Anesth Reanim. 2011 Oct;30(10):764-5. doi: 10.1016/j.annfar.2011.06.006. Epub 2011 Jul 20. No abstract available. French. PMID 21764543
- [Background] 8. Australasian Society of Clinical Immunology and Allergy. Operating suite guidelines for latex allergic patients. [Available online from: www.allergy.org] accessed 15/08/2015.
- [Background] Binkley HM, Schroyer T, Catalfano J. Latex allergies: a review of recognition, evaluation, management, prevention, education, and alternative product use. J Athl Train. 2003 Apr;38(2):133-40. PMID 16558678
- See also: Website of the Association of Surgical Technicians: Guideline statements for the Natural Rubber Latex Protein allergic patient in the operating room environment(adopted BOD October 2005, updated BOD January 2014). — http://www.ast.org
- See also: Website of the American Association of Nurse Anesthetists: Latex allergy management( Guidelines) — http://www.aana.org